CLINICAL TRIAL: NCT01896128
Title: Use of a Wakefulness-Promoting Agent (Armodafinil) Combined With Neuro-rehabilitation to Improve Neurological Recovery and to Reduce the Incidence of Disability in Patients Who Suffered a Stroke
Brief Title: Combining Armodafinil With Neuro-rehabilitation to Improve Neurological Recovery and Reduce Disability Post-Stroke
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Burke Rehabilitation Hospital (Other)
Collaborators: Teva Branded Pharmaceutical Products R&D, Inc. (Industry)
Responsible Party: Principal Investigator, Pasquale Fonzetti, MD, PhD, Associate Director, Memory Evaluation and Treatment Service, Burke Rehabilitation Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: BRC-394
Record Dates: First submitted 2013-07-02; First posted 2013-07-11 (Estimated); Results first posted 2019-11-04 (Actual); Last update posted 2019-11-04 (Actual); Status verified 2019-10

CONDITIONS: Stroke; Cerebrovascular Accident; Hemiparesis
Keywords: stroke; CVA; cerebrovascular accident; hemiparesis; impairment; motor recovery; neuroplasticity; nuvigil; armodafinil
MeSH Terms: conditions — Stroke; Paresis | interventions — Modafinil

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Armodafinil (Experimental): 150 mg armodafinil administered 2 hours prior to start of therapeutic regimen for 10 consecutive days
  Interventions: Drug: Armodafinil
- Placebo (Placebo Comparator): inactive agent administered 2 hours prior to start of therapeutic regimen for 10 consecutive days
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Armodafinil
  Other Names: Nuvigil
  Arms: Armodafinil
Drug: Placebo — inactive pill manufactured to mimic Armodafinil 150 mg tablet
  Arms: Placebo

SUMMARY:
Armodafinil is an FDA approved medication with wakefulness-promoting properties. It is a relatively safe agent with interesting neurochemical effects on the catecholamine system, producing an improvement in cognitive function, particularly working memory in humans. When combined with intensive task-related training, armodafinil may accelerate motor recovery in chronic stroke patients.

The primary aim of this study is to determine whether administration of armodafinil during subacute post-stroke rehabilitation will augment cortical plasticity and enhance motor recovery. The primary hypothesis suggests that cortical plasticity will be enhanced by armodafinil and, therefore, will induce an improvement in motor function and better performances on measures of motor control.

ELIGIBILITY:
Inclusion Criteria:

* First clinical stroke, either cerebral infarction or intracerebral hemorrhage
* Severe hemiparesis as measured by a Fugl-Meyer motor scale score of 0-25
* Screening Motricity Index score of 0-83
* Date of stroke onset between 7 to 21 days prior to study inclusion

Exclusion Criteria:

* Age less than 18
* Previous clinical stroke
* Pregnant and/or nursing patients
* Major psychiatric history, including psychosis and history of substance abuse
* Dementia
* Known CNS pathology such as brain tumor
* Significant language dysfunction or severe neglect that hinders comprehension, participation, and barrier to testing
* Seizures
* Left ventricular hypertrophy (LVH)
* Mitral valve prolapse (MVP)
* Severe chronic renal failure or severe hepatic failure
* History or current use of anti-epileptic medications, psychostimulants, or neuroleptics
* Current use of diazepam, phenytoin, propranolol, tricyclic antidepressants, steroidal contraceptives, cyclosporine, or theophylline

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2008-01; Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pasquale Fonzetti, MD, PhD, Principal Investigator — The Burke Rehabilitation Hospital
Locations (1):
- The Burke Rehabilitation Hospital, White Plains, New York, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Armodafinil: 150 mg armodafinil administered 2 hours prior to start of therapeutic regimen for 10 consecutive days
  Armodafinil
Period: Overall Study
Arm/Group | Armodafinil | Placebo
Started | 8 | 11
Completed | 5 | 8
Not Completed | 3 | 3
Not completed — Withdrawal by Subject | 3 | 3

BASELINE CHARACTERISTICS:
Population: Of a total 19 subjects enrolled: 8 subjects were randomly allocated to the Armodafinil arm and 11 subjects to the placebo arm.
  Three subjects for each arm of the study withdrew from the study. At day 100, there were 5 subjects of the Armodafinil group and 8 subjects of the placebo group that completed the study
Groups:
- Total: Total of all reporting groups
Arm/Group | Armodafinil | Placebo | Total
Number analyzed (Participants) | 8 | 11 | 19
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 6 | 5 | 11
  >=65 years | 2 | 6 | 8
Age, Continuous [Mean (Standard Deviation); unit: years] | 65.4 (12.4) | 67.5 (9.5) | 66.45 (10.95)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 6 | 9
  Male | 5 | 5 | 10
Region of Enrollment [Number; unit: participants]
  United States | 8 | 11 | 19

OUTCOME MEASURES:

1. Primary Outcome: Change in Fugl-Meyer Assessment of Sensorimotor Function From Baseline to Day 100
Description: Fugl-Meyer Assessment (FMA) scale is an index to assess the sensorimotor impairment in individuals who have had a stroke.The maximum possible score in Fugl-Meyer scale is 226, which corresponds to full sensory-motor recovery. The Fugl-Meyer Assessment scale is an ordinal scale that has 3 points for each item. A zero score is given for the item if the subject cannot do the task. A score of 1 is given when the task is performed partially and a score of 2 is given when the task is performed fully. However, reflex activity is measured using 2 points only, with a score of 0 or 2 for absence and presence of reflex respectively. The five domains assessed by Fugl-Meyer scale are:
  * Motor function (Maximum score in upper limb = 66;Maximum score in lower limb = 34)
  * Sensory function (Maximum score = 24)
  * Balance (Maximum score = 14)
  * Range of motion of joints (Maximum score = 44)
  * Joint pain (Maximum score = 44)
Time Frame: Baseline to Day 100
Population: data available for participants who completed the study
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Armodafinil | Placebo
Number analyzed (Participants) | 5 | 8
units on a scale
  Baseline | 14.8 (8.6) | 12.8 (7.0)
  Day100 | 39.7 (15.0) | 37.8 (20.9)

2. Secondary Outcome: Change in Functional Independence Measure (FIM) From Baseline to Day 100
Description: The FIM is used by health care practitioners to assess and grade the functional status of a person based on the level of assistance he or she requires.
  The motor subscale includes:Eating,Grooming,BathingDressing, upper body,Dressing, lower body Toileting Bladder management Bowel management Transfers - bed/chair/wheelchairTransfers - toiletTransfers - bath/showerWalk/wheelchairStairs The cognition subscale includes:Comprehension ExpressionSocial interaction Problem solvingMemory Each item is scored on a 7 point ordinal scale, ranging from a score of 1(worse) to a score of 7(better). The total score for the FIM motor subscale (the sum of motor subscale ) will be a value between 13 and 91.The total score for the FIM cognition subscale (the sum of the individual cognition subscale items) will be a value between 5(worse outcome) & 35(best outcome).The total score for the FIM instrument (the sum of subscale scores) will be a value between 18(worse outcome) & 126 (best outcome)
Time Frame: Day 100
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Armodafinil | Placebo
Number analyzed (Participants) | 8 | 11
units on a scale
  Baseline | 55.5 (17.8) | 52.4 (14.5)
  Day100 | 89.2 (21.7) | 90.9 (17.4)

3. Secondary Outcome: Timed 3-Minute Walk Test From Baseline to Day 100
Description: The 3MWT is a simple measure of the distance a person can walk in three minutes. Rest breaks are allowed if needed. The person is encouraged to walk as fast as they can, safely, for two minutes. Walking aids can be used as needed e.g. for elderly people with a record made of walking aid used.A clear course such as a hallway with cones or similar to mark an approximately 15m "out and back" course[8], stopwatch, pen and paper or a device to record distance walked.
Time Frame: Day 1, Day 100
Measure: Mean (Standard Deviation); unit: feet
Arm/Group | Armodafinil | Placebo
Number analyzed (Participants) | 8 | 11
feet
  Baseline | 49.4 (43.5) | 152.5 (89.2)
  Day100 | 152.5 (89.2) | 103.3 (73.8)

4. Secondary Outcome: NIH Stroke Scale (NIHSS)
Description: The National Institutes of Health Stroke Scale, or NIH Stroke Scale (NIHSS) is a tool used by healthcare providers to objectively quantify the impairment caused by a stroke. The NIHSS is composed of 11 items, each of which scores a specific ability between a 0 and 4. For each item, a score of 0 typically indicates normal function in that specific ability, while a higher score is indicative of some level of impairment. The individual scores from each item are summed in order to calculate a patient's total NIHSS score. The maximum possible score is 42, with the minimum score being a 0 Score.
  Stroke severity 0 No stroke symptoms 1-4 Minor stroke 5-15 Moderate stroke 16-20 Moderate to severe stroke 21-42 Severe stroke
Time Frame: Baseline Day 100
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Armodafinil | Placebo
Number analyzed (Participants) | 8 | 11
units on a scale
  Baseline | 11.9 (3.9) | 13.4 (3.3)
  Day100 | 6.7 (2.5) | 7.3 (2.7)

5. Secondary Outcome: 9-Hole Peg Test
Description: 9 HOLE PEG TEST
  * Administered by asking the client to take the pegs from a container, one by one, and place them into the holes on the board, as quickly as possible
  * Participants must then remove the pegs from the holes, one by one, and replace them back into the container
  * The board should be placed at the client's midline, with the container holding the pegs oriented towards the hand being tested
  * Only the hand being evaluated should perform the test
  * Hand not being evaluated is permitted to hold the edge of the board in order to provide stability
  * Scores are based on the time taken to complete the test activity, recorded in seconds
  * Alternative scoring - the number of pegs placed in 50 or 100 seconds can be recorded. In this case, results are expressed as the number of pegs placed per second
  * Stopwatch should be started from the moment the participant touches the first peg until the moment the last peg hits the container
Time Frame: Baseline & Day 100
Measure: Mean (Standard Error); unit: Seconds
Arm/Group | Armodafinil | Placebo
Number analyzed (Participants) | 8 | 11
Seconds
  Baseline | 34.0 (8.8) | 34.2 (9.5)
  Day100 | 27.3 (6.7) | 29.7 (6.1)

ADVERSE EVENTS:
Time Frame: 100 days
Arm/Group | Armodafinil | Placebo
All-Cause Mortality (participants affected / at risk) | 0/8 | 0/11
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/11
Other Adverse Events (participants affected / at risk) | 1/8 | 0/11
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Armodafinil (N=8) | Placebo (N=11)
Nervesousness (Nervous system disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No